CLINICAL TRIAL: NCT03531905
Title: A Randomized Study to Evaluate the Efficacy and Safety of Bempedoic Acid 180 + Ezetimibe 10 Fixed-Dose Combination Compared to Ezetimibe and Placebo In Subjects With T2DM and Elevated LDL-Cholesterol
Brief Title: Bempedoic Acid + Ezetimibe Fixed-Dose Combination (FDC) Study in Patients With Type 2 Diabetes and Elevated LDL-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002FDC-058
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Cholesterolemia
Keywords: diabetes; cholesterolemia; type 2 diabetes; LDL-C; T2D; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bempedoic acid + Ezetimibe FDC (Experimental): Bempedoic acid + Ezetimibe FDC Oral Tablet; Placebo oral capsule
  Interventions: Drug: Bempedoic acid + Ezetimibe FDC Oral Tablet; Drug: Placebo oral capsule
- Ezetimibe 10 mg (Active Comparator): Ezetimibe 10Mg Oral Tablet; Placebo Oral Tablet
  Interventions: Drug: Ezetimibe 10 mg Oral Tablet; Drug: Placebo Oral Tablet
- Placebo (Placebo Comparator): Placebo Oral Tablet, Placebo oral capsule
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Bempedoic acid + Ezetimibe FDC Oral Tablet — Experimental therapy of bempedoic acid 180 mg + ezetimibe 10 mg FDC tablet
  Arms: Bempedoic acid + Ezetimibe FDC
Drug: Ezetimibe 10 mg Oral Tablet — Ezetimibe 10 mg tablet, overencapsulated for blinding purposes
  Other Names: Zetia
  Arms: Ezetimibe 10 mg
Drug: Placebo Oral Tablet — Placebo tablet, matched for the FDC product for blinding purposes
  Arms: Ezetimibe 10 mg; Placebo
Drug: Placebo oral capsule — Placebo over-encapsulated for blinding purposes
  Arms: Bempedoic acid + Ezetimibe FDC; Placebo

SUMMARY:
12 week study to assess the LDL-C lowering efficacy, other lipid and glycemic measures, and safety of bempedoic acid/ezetimibe FDC compared to ezetimibe and placebo in patients with type 2 diabetes (T2D) and elevated LDL-C

DETAILED DESCRIPTION:
Assess efficacy of FDC vs. ezetimibe vs. placebo for 12 week LDL-C lowering, changes in atherogenic lipids, hsCRP and exploratory glycemic measures as well as safety in patients with type 2 diabetes and elevated LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for 6 months or greater
* Currently taking stable diabetes medication for 3 months or greater
* HbA1c between 7-10%
* LDL-cholesterol greater than 70 mg/dL
* Women must not be pregnant, lactating, or planning to become pregnant within 30 days after last dose of study medication; and must be postmenopausal, surgically sterile, or willing to use 1 acceptable form of birth control during the study through 30 days after the last dose of study medication

Exclusion Criteria:

* Body mass index > 40 kg/m2
* History of documented clinically significant cardiovascular disease
* Fasting triglycerides > 400 mg/dL
* History of Type 1 diabetes
* Uncontrolled hypothyroidism, liver dysfunction, renal dysfunction, gastrointestinal condition that may affect drug absorption, hematologic or coagulation disorder or active malignancy
* History of drug or alcohol abuse within 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (4):
- United States (4):
  - Clinical Trials Research, Lincoln, California
  - FInlay Medical Research, Miami, Florida
  - L-MARC Research Center, Louisville, Kentucky
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236

RESULTS

PARTICIPANT FLOW:
Groups:
- Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC: Participants received bempedoic acid + ezetimibe fixed-dose combination (FDC) 180 milligrams (mg)/10 mg tablets orally once daily for 12 weeks.
- Ezetimibe 10 mg: Participants received ezetimibe 10 mg overencapsulated tablets orally once daily for 12 weeks.
- Placebo: Participants received placebo to match the FDC 180 mg/10 mg tablet or the ezetimibe 10 mg overencapsulated tablet, taken orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Started | 81 | 81 | 80
Completed | 74 | 76 | 77
Not Completed | 7 | 5 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Participant was out of town | 1 | 0 | 0
Not completed — Could not speak with the participant | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo | Total
Number analyzed (Participants) | 81 | 81 | 80 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.65) | 61.0 (8.00) | 62.1 (8.63) | 61.4 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 42 | 117
  Male | 45 | 42 | 38 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 38 | 30 | 100
  Not Hispanic or Latino | 49 | 43 | 50 | 142
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 15 | 16 | 46
  White | 61 | 65 | 62 | 188
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the average of Screening Visit 3 (Visit S3) and Treatment Visit 1 (Visit T1) values (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Population: Efficacy Analysis Set: all randomized participants who received at least one dose of investigational medicinal product (Full Analysis Set), excluding participants at 3 study sites
  milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 145.06 (31.504) | 139.24 (28.121) | 143.36 (26.421) | 142.55 (28.715)
High-sensitivity C-reactive protein (hsCRP) [Median (Inter-Quartile Range); unit: milligrams per liter (mg/ L)] — Baseline was defined as the last value prior to the first dose of investigational medicinal product (IMP). Population: Efficacy Analysis Set
  milligrams per liter (mg/ L)
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 2.570 [1.735 to 4.860] | 2.420 [1.545 to 5.590] | 3.480 [1.520 to 8.040] | 2.610 [1.550 to 5.740]
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the average of Visit S3 and Visit T1 values (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 181.69 (36.659) | 172.87 (33.277) | 177.38 (29.116) | 177.31 (33.194)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the average of Visit S3 and Visit T1 values (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 230.34 (37.234) | 221.33 (33.592) | 225.94 (32.830) | 225.87 (34.619)
Apolipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last value prior to the first dose of IMP. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 121.6 (22.95) | 117.3 (22.96) | 120.8 (18.53) | 119.9 (21.56)
Triglycerides (TGs) [Median (Inter-Quartile Range); unit: mg/dL] — Baseline was defined as the average of Visit S3 and Visit T1 values (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 172.25 [127.50 to 238.50] | 159.25 [118.25 to 236.50] | 163.00 [124.50 to 219.50] | 163.00 [121.00 to 232.50]
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the average of Visit S3 and Visit T1 values (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 48.73 (13.067) | 47.95 (10.847) | 48.53 (13.482) | 48.40 (12.447)
Hemoglobin A1C (HbA1c) [Mean (Standard Deviation); unit: Percent] — Baseline was defined as the last value prior to the first dose of IMP. Population: Efficacy Analysis Set
  Percent
    number analyzed (Participants) | 60 | 60 | 59 | 179
    (all) | 7.86 (0.927) | 7.96 (1.279) | 8.02 (0.773) | 7.95 (1.013)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last value prior to the first dose of IMP. Population: Efficacy Analysis Set
  mg/dL
    number analyzed (Participants) | 58 | 58 | 57 | 173
    (all) | 162.4 (46.10) | 153.3 (46.73) | 174.2 (57.53) | 163.2 (50.78)
HOMA-IR index [Mean (Standard Deviation); unit: units on a scale] — Baseline was defined as the last value prior to the first dose of study drug (on or before T1). Normal HOMA-IR values range from 0.5 to 1.4. A value less than 1.0 indicates insulin sensitivity. A value above 1.9 indicates early insulin resistance. A value above 2.9 indicates significant insulin resistance. A higher number indicates increased insulin resistance. Population: Efficacy Analysis Set
  units on a scale
    number analyzed (Participants) | 57 | 56 | 53 | 166
    (all) | 6.709 (6.200) | 10.847 (18.074) | 13.267 (21.305) | 10.199 (16.503)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12/End of Study (EOS) in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the average of LDL-C values at the Screening Visit 3 (Visit S3) and the Treatment Visit 1 (Visit T1) (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for LDL-C was analyzed using analysis of covariance (ANCOVA), with treatment as factor and Baseline lipid parameter as a covariate. Missing data for LDL-C was imputed using the last observation carried forward (LOCF) method. Percent change from Baseline was calculated as: ([LDL-C value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For LDL-C, if a measured LDL-C value was available, measured LDL-C was used.
Time Frame: Baseline; Week 12
Population: Efficacy Analysis Set (EAS): all randomized participants who received at least one dose of investigational medicinal product (Full Analysis Set), excluding participants at three study sites. Only participants with available data were analyzed.
Measure: Geometric Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 59 | 57
Percent change | -38.8 (2.24) | -19.2 (2.16) | 0.9 (2.20)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of Least Squares (LS) means = -39.6, 95% CI 2-sided [-45.8 to -33.4], Standard Error of Mean 3.14
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -19.5, 95% CI 2-sided [-25.7 to -13.4], Standard Error of Mean 3.11
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -20.1, 95% CI 2-sided [-26.2 to -14.0], Standard Error of Mean 3.08

2. Secondary Outcome: Percent Change From Baseline to Week 12/EOS in LDL-C (Comparing Ezetimibe With Placebo)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the average of LDL-C values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for LDL-C was analyzed using ANCOVA, with treatment as factor and Baseline lipid parameter as a covariate. Missing data for LDL-C was imputed using the LOCF method. Percent change from Baseline was calculated as: ([LDL-C value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For LDL-C, if a measured LDL-C value was available, measured LDL-C was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 59 | 57
Percent change | -19.2 (2.16) | 0.9 (2.20)
Statistical Analysis 1: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -20.1, 95% CI 2-sided [-26.2 to -14.0], Standard Error of Mean 3.08

3. Secondary Outcome: Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for hsCRP. Baseline was defined as the last value prior to the first dose of investigational medicinal product (IMP). Percent change from Baseline for hsCRP was analyzed using a non-parametric approach. Percent change from Baseline was calculated as: ([hsCRP value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For hsCRP, if a measured hsCRP value was available, measured hsCRP was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
Percent change | -25.347 [-48.980 to 3.292] | 2.078 [-22.610 to 48.770] | 14.085 [-21.642 to 50.776]
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank sum test; Location shift = -36.7, 95% CI 2-sided [-55.97 to -17.67], Standard Error of Mean 9.77
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.005, Wilcoxon rank sum test; Location shift = -29.2, 95% CI 2-sided [-48.92 to -9.62], Standard Error of Mean 10.03
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.480, Wilcoxon rank sum test; Location shift = -7.5, 95% CI 2-sided [-30.51 to 13.76], Standard Error of Mean 11.29

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for non-HDL-C. Baseline was defined as the average of non-HDL-C values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for non-HDL-C was analyzed using ANCOVA, with treatment as factor and Baseline lipid parameter as a covariate. Missing data for non-HDL-C was imputed using the LOCF method. Percent change from Baseline was calculated as: ([non-HDL-C value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For non-HDL-C, if a measured non-HDL-C value was available, measured non-HDL-C was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 59 | 57
Percent change | -33.0 (2.01) | -17.8 (1.94) | 0.1 (1.97)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -33.1, 95% CI 2-sided [-38.6 to -27.5], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -15.3, 95% CI 2-sided [-20.8 to -9.7], Standard Error of Mean 2.80
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -17.8, 95% CI 2-sided [-23.3 to -12.4], Standard Error of Mean 2.76

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the average of TC values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for TC was analyzed using ANCOVA, with treatment as factor and Baseline lipid parameter as a covariate. Missing data for TC was imputed using the LOCF method. Percent change from Baseline was calculated as: ([TC value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For TC, if a measured TC value was available, measured TC was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 59 | 57
Percent change | -27.3 (1.61) | -13.9 (1.55) | -0.1 (1.57)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -27.2, 95% CI 2-sided [-31.7 to -22.8], Standard Error of Mean 2.25
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -13.4, 95% CI 2-sided [-17.8 to -9.0], Standard Error of Mean 2.24
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -13.9, 95% CI 2-sided [-18.2 to -9.5], Standard Error of Mean 2.21

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (Apo B)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for apo B. Baseline was defined as the last value prior to the first dose of IMP. Percent change from Baseline for TC was analyzed using ANCOVA, with treatment as factor and Baseline lipid parameter as a covariate. Missing data for apo B was imputed using the LOCF method. Percent change from Baseline was calculated as: ([apo B value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For apo B, if a measured apo B value was available, measured apo B was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 59 | 57
Percent change | -27.5 (1.94) | -14.8 (1.88) | -0.3 (1.91)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -27.2, 95% CI 2-sided [-32.6 to -21.8], Standard Error of Mean 2.73
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -12.8, 95% CI 2-sided [-18.1 to -7.4], Standard Error of Mean 2.71
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -14.4, 95% CI 2-sided [-19.7 to -9.1], Standard Error of Mean 2.68

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Triglycerides (TGs)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for TGs. Baseline was defined as the average of TG values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for TGs was analyzed using a non-parametric approach. Percent change from Baseline was calculated as: ([TG value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For TGs, if a measured TG value was available, measured TG was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
Percent change | -9.20 [-27.97 to 19.39] | -13.59 [-28.58 to 1.33] | -5.11 [-19.84 to 12.15]
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p = 0.457, Wilcoxon rank sum test; Location shift = -3.9, 95% CI 2-sided [-14.55 to 6.79], Standard Error of Mean 5.44
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.351, ANCOVA; Difference of LS means = 4.7, 95% CI 2-sided [-4.93 to 15.63], Standard Error of Mean 5.25
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.068, ANCOVA; Difference of LS means = -9.2, 95% CI 2-sided [-17.92 to 0.68], Standard Error of Mean 4.75

8. Secondary Outcome: Percent Change From Baseline to Week 12 in High-density Lipoprotein Cholesterol (HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for HDL-C. Baseline was defined as the average of HDL-C values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. Percent change from Baseline for HDL-C was analyzed using ANCOVA, with treatment as factor and Baseline lipid parameter as a covariate. Missing data for HDL-C was imputed using the LOCF method. Percent change from Baseline was calculated as: ([HDL-C value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For HDL-C, if a measured HDL-C value was available, measured HDL-C was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 59 | 57
Percent change | -5.1 (1.53) | 2.1 (1.48) | 0.8 (1.50)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p = 0.007, ANCOVA; Difference of LS means = -5.9, 95% CI 2-sided [-10.1 to -1.7], Standard Error of Mean 2.14
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -7.3, 95% CI 2-sided [-11.5 to -3.1], Standard Error of Mean 2.12
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.517, ANCOVA; Difference of LS means = 1.4, 95% CI 2-sided [-2.8 to 5.5], Standard Error of Mean 2.11

9. Secondary Outcome: Number of Participants With LDL-C <70 Milligrams Per Deciliter (mg/dL) at Week 12
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for LDL-C. For LDL-C, if a measured LDL-C value was available, measured LDL-C was used.
Time Frame: Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
Participants | 21 | 3 | 0
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.118, Fisher Exact
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, Fisher Exact

10. Secondary Outcome: Secondary Outcome Measure: Number of Participants With an LDL-C Reduction of ≥50% From Baseline at Week 12
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the average of LDL-C values at Visit S3 and Visit T1 (last 2 non-missing values on or prior to Day 1). If only 1 value was available, the single value was used as Baseline. LDL-C reduction from Baseline was calculated as the LDL-C value at Week 12 minus the Baseline value. For LDL-C, if a measured LDL-C value was available, measured LDL-C was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
Participants | 22 | 0 | 0
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, Fisher Exact

11. Secondary Outcome: Change From Baseline to Week 12 in Hemoglobin A1C (HbA1c)
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for HbA1c. Baseline was defined as the last value prior to the first dose of IMP (on or before Visit T1). Change from Baseline was calculated as the HbA1c value at Week 12 minus the Baseline value. For HbA1c, if a measured HbA1c value was available, measured HbA1c was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
mg/dL | 0.01 (0.849) | -0.06 (0.851) | 0.03 (0.667)

12. Secondary Outcome: Percent Change From Baseline to Week 12 in HbA1c
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for HbA1c. Baseline was defined as the last value prior to the first dose of IMP (on or before Visit T1). Percent change from Baseline for HbA1C was analyzed using ANCOVA, with treatment as factor and Baseline HbA1C value as a covariate. Percent change from Baseline for HbA1c was calculated as: ([HbA1c value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For HbA1c, if a measured HbA1c value was available, measured HbA1c was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 54 | 56 | 57
Percent change | 0.1 (1.31) | -0.7 (1.28) | 0.4 (1.27)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p = 0.877, ANCOVA; Difference of LS means = -0.3, 95% CI 2-sided [-3.9 to 3.3], Standard Error of Mean 1.83
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.669, ANCOVA; Difference of LS means = 0.8, 95% CI 2-sided [-2.8 to 4.4], Standard Error of Mean 1.83
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.556, ANCOVA; Difference of LS means = -1.1, 95% CI 2-sided [-4.6 to 2.5], Standard Error of Mean 1.81

13. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Fasting Plasma Glucose
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Samples were collected and analyzed for fasting plasma glucose. Baseline was defined as the last value prior to the first dose of study drug (on or before T1). Percent change from Baseline for fasting plasma glucose was analyzed using ANCOVA, with treatment as factor and Baseline fasting plasma glucose as a covariate. Percent change from Baseline for fasting plasma glucose was calculated as: ([fasting plasma glucose value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For fasting plasma glucose, if a measured fasting plasma glucose value was available, measured fasting plasma glucose was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 53 | 55 | 55
Percent change | 4.2 (3.29) | 3.7 (3.28) | 1.7 (3.27)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p = 0.589, ANCOVA; Difference of LS means = 2.5, 95% CI 2-sided [-6.7 to 11.7], Standard Error of Mean 4.64
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.904, ANCOVA; Difference of LS means = 0.6, 95% CI 2-sided [-8.6 to 9.7], Standard Error of Mean 4.64
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.676, ANCOVA; Difference of LS means = 2.0, 95% CI 2-sided [-7.3 to 11.2], Standard Error of Mean 4.66

14. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in 2-hour Post Prandial Plasma Glucose (PPG)
Description: Blood samples were drawn 2 hours ± 5 minutes after the start of the meal. Samples were collected and analyzed for PPG. Baseline was defined as the last value prior to the first dose of study drug (on or before T1). Percent change from Baseline for PPG was calculated as: ([PPG value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100. For PPG, if a measured PPG value was available, measured PPG was used.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 55 | 53 | 50
Percent change | 1.9 (24.25) | 0.2 (31.88) | 2.2 (25.39)

15. Other Pre Specified Outcome: Percent Change From Baseline to Week 12 in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) Index
Description: The HOMA-IR index was calculated from the fasting glucose and insulin values that were obtained at each clinic visit (Day 1/Visit T1, Week 4/Visit T2, and Week 12/Visit T3) during the double-blind treatment period, using the formula: (fasting glucose [millimoles per milliliter {mmol/ml}] x fasting insulin [micro International Units per milliliter {μIU/ml}]) divided by 22.5. Percent change from Baseline for HOMA-IR index was analyzed using ANCOVA, with treatment as factor and Baseline HOMA-IR index as a covariate. Baseline was defined as the last value prior to the first dose of study drug (on or before T1). Percent change from Baseline for HOMA-IR index was calculated as: ([HOMA-IR index value at Week 12 minus Baseline value] divided by [Baseline value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: EAS. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 51 | 53 | 55
Percent change | 3.0 (9.85) | 2.5 (9.59) | 18.9 (9.79)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p = 0.258, ANCOVA; Difference of LS means = -15.8, 95% CI 2-sided [-43.4 to 11.7], Standard Error of Mean 13.95
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.972, ANCOVA; Difference of LS means = 0.5, 95% CI 2-sided [-26.8 to 27.7], Standard Error of Mean 13.79
Statistical Analysis 3: Comparison: Ezetimibe 10 mg vs Placebo; Test type: Superiority; p = 0.235, ANCOVA; Difference of LS means = -16.3, 95% CI 2-sided [-43.3 to 10.7], Standard Error of Mean 13.68

16. Other Pre Specified Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) that began or worsened in severity on or after the first dose of double-blind IMP through 30 days after the last dose of double-blind IMP. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, including control, and which does not necessarily have a causal relationship with treatment. An AE is: any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product; any new disease or exacerbation of an existing disease; any deterioration in non-protocol-required measurements of a laboratory value or other clinical test (e.g., electrocardiogram or x-ray) that results in symptoms, a change in treatment, or discontinuation from IMP; or an adverse drug reaction.
Time Frame: up to approximately 16 weeks
Population: Safety Analysis Set: all randomized participants who received at least one dose of IMP
Measure: Count of Participants; unit: Participants
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 81 | 81 | 80
Participants | 55 | 45 | 46

ADVERSE EVENTS:
Time Frame: up to approximately 16 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began or worsened in severity on or after the first dose of double-blind investigational medicinal product (IMP) through 30 days after the last dose of double-blind IMP, were collected in members of the Safety Population (all randomized participants who received at least 1 dose of blinded IMP).
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Ezetimibe 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/81 | 1/81 | 1/80
Other Adverse Events (participants affected / at risk) | 8/81 | 6/81 | 7/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC (N=81) | Ezetimibe 10 mg (N=81) | Placebo (N=80)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC (N=81) | Ezetimibe 10 mg (N=81) | Placebo (N=80)
Bronchitis (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 3
Blood glucose increased (Investigations) | 3 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 2 | 1 | 4

LIMITATIONS AND CAVEATS:
Sites 5801003, 5801041, and 5801043 were suspected of Good Clinical Practice violations in an earlier Phase 3 trial (NCT03337308), hence the Efficacy Analysis Set (which excluded these 3 sites) was designated as the primary efficacy analysis set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03531905/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03531905/SAP_001.pdf